CLINICAL TRIAL: NCT01750944
Title: Validation of the Measurement of a Systolic Pressure Index at the Toe (IPSO) After a Walking Test
Brief Title: Measurement of a Systolic Pressure Index at the Toe After a Walking Test
Acronym: IPSO FACTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2012/APM-02; 2012-A01432-41 (Other: RCB number)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Good Health
Keywords: Blood pressure site; Good health; Brachial blood pressure; Ankle; Toe; Walking test; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers 1 (Experimental): The study population consists of adult, healthy volunteers randomized into two identical groups.
  Intervention: ankle first
  Interventions: Procedure: Ankle first
- Healthy Volunteers 2 (Experimental): The study population consists of adult, healthy volunteers randomized into two identical groups.
  Intervention: toe first
  Interventions: Procedure: Toe first

INTERVENTIONS:
Procedure: Ankle first — 1. Brachial blood pressure on both the left and right (BBP-LR) sides is measured, as well as at the left and right ankles (BPA-LR).
  2. A 15 minute walking test (WT) is performed.
  3. BBP-LR and BPA-LR are re-measured.
  4. 2 hours of rest.
  5. BBP-LR and the blood pressure at the left and right big toes (BPT-LR) are measured.
  6. WT is reperformed.
  7. BBP-LR and BPT-LR are re-measured.
  Arms: Healthy Volunteers 1
Procedure: Toe first — 1. Brachial blood pressure on both the left and right (BBP-LR) sides is measured, as well as at the left and right big toes (BPT-LR).
  2. A 15 minute walking test (WT) is performed.
  3. BBP-LR and BPT-LR are re-measured.
  4. 2 hours of rest.
  5. BBP-LR and the blood pressure at the left and right ankles (BPA-LR) are measured.
  6. WT is reperformed.
  7. BBP-LR and BPA-LR are re-measured.
  Arms: Healthy Volunteers 2

SUMMARY:
The main objective of this study is to evaluate the concordance of the variation in systolic pressure indices measured at the toe and ankle after a walking test in healthy volunteers.

DETAILED DESCRIPTION:
Our secondary objectives are:

* to evaluate the concordance between left- and right-side measures: systolic pressure indices measured at the toe after a walking test (healthy volunteers)
* to evaluate the concordance between left- and right-side measures: systolic pressure indices measured at the ankle after a walking test (healthy volunteers)
* to evaluate the concordance of the variation in systolic pressure indices measured at the toe and ankle during the recuperation phase after a walking test (5 and 10 minutes after end of walking test) in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* The subject must have given his/her informed and signed consent
* The subject must be insured or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is in an exclusion period determined by a previous study
* The subject is under judicial protection, under tutorship or curatorship
* The subject refuses to sign the consent
* It is impossible to correctly inform the subject
* The subject is pregnant, parturient, or breastfeeding
* The subject has a contraindication for a walking test
* Presence of mediacalcose objectified by a Doppler examination of the anterior and posterior tibial arteries, performed on the test day
* Known history of cardiovascular disease
* Poorly controlled diabetes or hypertension
* Neurological, muscular or rheumatic pathology contra-indicating a walking test
* Acute transient infection (cold-rhinitis, flu, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Difference between brachial and ankle blood pressure | Before effort test (minute -15, day 0)
Difference between brachial and ankle blood pressure | After effort test (minute 0, day 0)
Difference between brachial and toe blood pressure | Before effort test (minute -15, day 0)
Difference between brachial and toe blood pressure | After effort test (minute 0, day 0)

SECONDARY OUTCOMES:
Brachial blood pressure, left arm | Before effort test (minute -15, day 0)
Brachial blood pressure, left arm | After effort test (minute 0, day 0)
Brachial blood pressure, left arm | After effort test (minute 5, day 0)
Brachial blood pressure, left arm | After effort test (minute 10, day 0)
Brachial blood pressure, right arm | Before effort test (minute -15, day 0)
Brachial blood pressure, right arm | After effort test (minute 0, day 0)
Brachial blood pressure, right arm | After effort test (minute 5, day 0)
Brachial blood pressure, right arm | After effort test (minute 10, day 0)
Blood pressure, left big toe | Before effort test (minute -15, day 0)
Blood pressure, left big toe | After effort test (minute 0, day 0)
Blood pressure, left big toe | After effort test (minute 5, day 0)
Blood pressure, left big toe | After effort test (minute 10, day 0)
Blood pressure, right big toe | Before effort test (minute -15, day 0)
Blood pressure, right big toe | After effort test (minute 0, day 0)
Blood pressure, right big toe | After effort test (minute 5, day 0)
Blood pressure, right big toe | After effort test (minute 10, day 0)
Blood pressure, right ankle | Before effort test (minute -15, day 0)
Blood pressure, right ankle | After effort test (minute 0, day 0)
Blood pressure, right ankle | After effort test (minute 5, day 0)
Blood pressure, right ankle | After effort test (minute 10, day 0)
Blood pressure, left ankle | Before effort test (minute -15, day 0)
Blood pressure, left ankle | After effort test (minute 0, day 0)
Blood pressure, left ankle | After effort test (minute 5, day 0)
Blood pressure, left ankle | After effort test (minute 10, day 0)

OTHER OUTCOMES:
Time at which the tests were performed (hh:mm) | Day 0
The volunteer is an athlete? yes/no | Day 0; baseline
The volunteer drank coffee before the test? yes/no | Day 0; baseline
The volunteer is a smoker? yes/no | Day 0; baseline
Description of treatments currently being taken | Day 0; baseline

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Perez Martin, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France